CLINICAL TRIAL: NCT02190734
Title: Inpatient Rehabilitation Treatments and Effect on Pushing Behaviors in Individuals Post-stroke
Brief Title: Pushing Behaviors in Individuals Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Thomas G Hornby, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pusher1
Record Dates: First submitted 2014-05-21; First posted 2014-07-15 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Stroke
Keywords: Stroke; Pusher Syndrome; Lateropulsion; Pushing Behaviors; Burke Lateropulsion Scale
MeSH Terms: conditions — Stroke | interventions — Sitting Position; Wheelchairs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- wheelchair, walking on treadmill, walking overground (Other): Sitting in wheel chair Gait training on treadmill Gait training overground
  Interventions: Other: Sitting in wheel chair; Other: Gait training on treadmill; Other: Gait training overground

INTERVENTIONS:
Other: Sitting in wheel chair — Placebo/control intervention- No treatment, sitting in a wheelchair for 30 minutes
Other: Gait training on treadmill — Walking on a treadmill with or without body weight support during 30 minute treatment
Other: Gait training overground — Walking overground with or without body weight support during 30 minute treatment

SUMMARY:
Some individuals demonstrate pushing behaviors after having a stroke. The purpose of this study is to see if there are immediate changes in pushing behaviors in individuals who have had a stroke before and after sitting in a wheelchair, walking on the treadmill, and walking overground.

The investigators do not think there will be a change with sitting in the wheelchair, but the investigators think there may be an improvement in pushing behaviors after walking training.

DETAILED DESCRIPTION:
The study population of interest is primarily individuals in inpatient rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* score >0 in each subsection of the Scale for Contraversive Pushing
* admitted to the Rehabilitation Institute of Chicago inpatient rehabilitation setting
* stroke within previous 180 days
* consent to participate in the study
* ambulating greater than 150' at a time prior to stroke

Exclusion Criteria:

* other neurologic diagnoses
* weight bearing precautions, orthopedic injuries, or other medical co-morbidities that prevent adherence to the study protocol

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Burke Lateropulsion Scale | Before and after each of 3 treatment sessions (3 separate days) over a maximum of a 10 day period
  Clinical measure of pushing behaviors in supine, sitting, standing, walking, and transfers will be performed before and after each 30 minute training session.

CONTACTS AND LOCATIONS:
Overall Officials: T. George Hornby, PT, PhD, Principal Investigator — Rehabilitation Institute of Chicago, University of Illinois at Chicago
Locations (2):
- United States (2):
  - Rehabilitation Hospital of the Pacific, Honolulu, Hawaii
  - Rehabilitation Institute of Chicago, Chicago, Illinois